CLINICAL TRIAL: NCT03468556
Title: A Randomized, Double-Blind, Placebo Controlled Study to Assess the Efficacy and Safety of SNP-610 for the Treatment of Patients With Non-alcoholic Steatohepatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNP-610-201
Record Dates: First submitted 2018-03-06; First posted 2018-03-16 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: test drug
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test drug (Experimental): 2 tabs of SNP-610
  Interventions: Drug: SNP-610
- placebo (Placebo Comparator): 2 tabs of placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: SNP-610 — Subjects will take 2 tablets once a day orally for 12 weeks
  Arms: test drug
Drug: Placebo Oral Tablet — Subjects will take 2 tablets once a day orally for 12 weeks
  Arms: placebo

SUMMARY:
The primary objective of the study is to compare the changes in serum ALT level among patients with non-alcoholic steatohepatitis (NASH) following 3-month treatment of 800 mg SNP-610 or the placebo. The secondary objectives will be to compare the changes in liver fat fraction, other liver function tests, cytokeratin-18 (CK-18) fragment level and adverse event / serious adverse event rates among the interventional and placebo arms.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo controlled study will be conducted in medical centers around Taiwan.

The objective of the study is to investigate the efficacy and safety of SNP-610 for the treatment of NASH, assuming the treatment efficacy of the investigational product is superior to the placebo control.

Subjects who fulfill all the entry criteria and have written informed consent will be enrolled to the study. Eligible subjects will be randomized in a 1:1 ratio to receive study drug or placebo control. Considering a 10% drop-out rate, approximately 80 subjects will be enrolled in order to recruit 70 evaluable subjects, each arm will be at least 35 evaluable subjects to complete the enrollment.

Subjects will be administered the test drugs or placebo oral daily for 3 months or until treatment terminates prematurely. Subjects will return to the study center for clinical evaluation once every 4 weeks throughout the treatment period. Clinical assessment procedures and laboratory tests including ultrasound imaging, hematology with differential, biochemistry, liver function panel, and urinalysis, will be performed at each study visit. The primary endpoint assessment will be the reduction of ALT at completion of Week 12 treatment.

Subjects who finish treatment or discontinue prematurely from the study for any reason after receiving one or more doses of study drug will be assessed for safety for 2 (±1) weeks after the last study drug dose or longer in the case of any significant AE or abnormal biochemical or clinical finding.

Each subject will participate in the study for approximately 14 weeks (including the enrollment/baseline visit, 3 routine monthly visits during treatment period, and 1 follow-up visit after 2 weeks of the end of treatment).

It is assumed the study will include a 6 months enrollment period and a further 4 months to complete the follow-up for all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Body weight ≥ 54 kg
3. Diagnosis of non-alcoholic steatohepatitis (NASH) as evidenced by imaging or other diagnostic assessments. Subject should have documented liver fat content ≥ 10.0 % as measured by MRI method prior to study drug administration.
4. Alanine aminotransferase (ALT) levels ≥ 2.0x upper limit of normal (ULN) on at least two occasions, seven or more days apart, prior to study drug administration
5. Have adequate organ functions as defined by the following examinations prior to the start of study treatment:

   1. Hematology: Hemoglobin ≥ 9 g/dL, a platelet count ≥ 100 x 10^9/L, and a white blood cell count ≥ 3.0 x 10^9/L
   2. Renal: creatinine clearance ≥ 90 mL/min (by Cockcroft-Gault equation), serum uric acid < 9.0 mg/dL
6. Able to provide written informed consent, and understand and comply with the requirements of the study

Exclusion Criteria:

1. Decompensated or severe liver disease as evidenced by one or more of the following:

   1. Confirmed cirrhosis or suspicion of cirrhosis
   2. Liver transplant
   3. Liver malignancy
   4. Ascites
   5. Bilirubin >2 x ULN, or ALT or AST > 10 x ULN
   6. Acute or chronic hepatitis A, B, C, HIV, or other liver diseases affecting liver function.

   Patients with cysts, hemangiomas, or similar abnormalities, are accepted.
2. History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120-mL wine or 14 cans of 350-mL beer), or other substance abuse within the prior two years
3. Subjects who are unable to undergo an MRI scan.
4. Subjects have electronically, magnetically and mechanically activated implanted devices, including but not limited to automatic cardioverter defibrillators, cardiac pacemakers, insulin pumps, metallic splinters in the eye, ferromagnetic haemostatic clips in central nervous systems or vascular vessels.
5. Significant systemic or major illness other than liver disease, including auto-immune disease, coronary artery disease, cerebrovascular disease, malignant neoplasms, pulmonary disease, renal insufficiency, serious psychiatric disease, and/or other serious disease, that, in the opinion of the Investigator would preclude the subject from participating in and completing the study
6. Documented history of serious allergic reaction to SNP-610 or any structurally related compounds
7. Diabetic patients who have not maintained a stable dose of oral medication for hyperglycemia or have had more than 10 percent change in their insulin dose over the past two months
8. Regular use of agents that are potent against hepatitis or affecting lipid metabolisms, including but not limited to HMGCoA reductase inhibitors (statins), fibrates, silymarin, N-acetylcysteine, or anti-TNF therapies.

   Note: refer to Section 6.5 Prohibited agents for details.
9. Pregnant or lactating
10. Female of child-bearing potential who are not committed to take reliable contraception during the participation of the study and at least 4 weeks after the end of the study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase | 12 weeks
  Absolute change from baseline in serum alanine aminotransferase (ALT/GPT)

SECONDARY OUTCOMES:
MRI liver FF | 12 weeks
  Absolute change from baseline in liver fat content
MRI liver FF | 12 weeks
  Relative change from baseline in liver fat content
Aspartate aminotransferase | 12 weeks
  Change in serum level at 12 weeks
Alkaline phosphatase | 12 weeks
  Change in serum level at 12 weeks
Gamma-glutamyl transpeptidase | 12 weeks
  Change in serum level at 12 weeks
Total bilirubin | 12 weeks
  Change in serum level at 12 weeks
Galactose single point | 12 weeks
  Change in serum level at 12 weeks
CK-18 | 12 weeks
  Change in serum level at 12 weeks

OTHER OUTCOMES:
Insulin resistance | 12 weeks
  Change in insulin resistance at Week 12
Triglycerides | 12 weeks
  Changes in serum at Week 12
Low density lipoprotein | 12 weeks
  Changes in serum at Week 12
Total cholesterol | 12 weeks
  Changes in serum at Week 12
High density lipoprotein | 12 weeks
  Changes in serum at Week 12
Gene expression biomarkers | 12 weeks
  Gene expression biomarkers (ACC1, Adfp, AOX, Cat, CCL20, CCR2, Cpt1α, CYP2E1, CYP4A11, CYP7A, Dgat1, Dgat2, FAS, Gapdh, Gpx1, Gpx2, Gpx3, Gpx4, GSS, Hadh, Ho1, HSL, IL-10, IL-1β, IL-6, iNOS, LCAD, NF-κB1, NF-κB2, Pparα, PPARβ/δ, PPARγ, SCD-1, Sod1, Sod2, Sod3, SREBP-1c, TGFβ, TLR4, TNFα, Ucp2, VLCAD, α-SMA, β-actin) related to NASH changes in blood at Week 12
Rate of patients who experience AEs leading to discontinuation at end of treatment | 12 weeks
Rate of patients who experience AE/SAE at end of treatment | 12 weeks

IPD SHARING:
Plan to Share IPD: Undecided